CLINICAL TRIAL: NCT06110052
Title: Clinical Presentations and Surgical Outcome of Obstructive Müllerian Anomalies: A Prospective Cohort Study
Brief Title: Clinical Presentations and Surgical Outcome of Obstructive Müllerian Anomalies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dina Ali Mahmoud Mohamed, Principal Investigator, Assiut University
Other Study IDs: OMAs
Record Dates: First submitted 2023-08-03; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Mullerian Duct Anomalies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: prospective follow up — compare preoperative and postoperative visual analog scale VAS of maximum perceived pain in ladies with OMAs

SUMMARY:
The present study aims at:

A. The main outcome is to compare preoperative and postoperative visual analog scale VAS from 0 to 10 of maximum perceived pain in ladies with OMAs.

1. description of clinical presentation and percentage of OMAs in relation to other Mullerian anomalies
2. description of different subtypes and its percentage.
3. description of the corrective procedures and their short-term outcomes.

DETAILED DESCRIPTION:
Obstructive Mullerian anomalies (OMAs) represent a real challenge in diagnosis and treatment, its incidence is not yet recognized. Care givers and gynecologist should be aware with its clinical presentation to avoid its delayed diagnosis and misdiagnosis. In addition, delayed diagnoses may result in retrograde menstruation, recurrent cyclic pains, chronic pelvic pains, poor quality of life and threats to future fertility.

Cases with complete obstructive Müllerian anomalies (C-OMAs) classically present with recurrent cyclic pains at puberty and their diagnosis is usually established easily. However, cases with Hemi obstructive anomalies (H-OMA) usually present with progressive dysmenorrhea and delayed diagnosis may result in pelvic adhesions, progressive hematosalpinx and endometriosis which directly threats natural future fertility. H-OMAs may results from obstructing uterine septa or unilateral cervical obstruction in a double uterus. Also, it may result from obstructing longitudinal vaginal septa in cases with double uterus, septate uterus or hybrid septate uterus .

A hybrid uterine anomaly is relatively a recent term that described the coexistence of septate and bicornuate uterus together. Pure septate uterus has a convex or flat fundus, when there is any fundal depression, it is termed hybrid septate uterus.

Pain with or without amenorrhoea is the main presentation of OMAs. Surgical correction should improve these symptoms. To the best of our knowledge there is no published prospective trials compared visual analog scale VAS in ladies with OMAs before and after surgical correction.

ELIGIBILITY:
Inclusion Criteria:

* All cases with OMAs or H-OMAs

Exclusion Criteria:

* Cases who refuse to participate in the study. 2.Cases who underwent previous surgical repair for their OMA or H-OMA.

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: demographic data will be collected about age, marital status, menarche, parity, consanguinity and family history.
  detailed history: about complaint and presenting symptoms will be obtained as delayed menarche, cyclic pain, abdominal distention, dull aching abdominal pain, dyspareunia and infertility physical examination:
  * general examination for secondary sexual characters, other anomalies
  * abdominal examination for abdominal mass, tenderness
  * genital examination by inspection for bulging hymen, per-vaginal examination
  * per- rectal examination investigation : CBC,, transvaginal, per-rectal, 3D abdominal ultrasonography
  Diagnosis:
  Anomalies will be categorized according to ESHRE classification 2016 Surgical procedure: follow up for the patient for three months for symptoms improvement and any complications.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
mullerian duct anomalies | 48 months
  A. The main outcome is to compare preoperative and postoperative visual analog scale VAS of maximum perceived pain in ladies with OMAs.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed F Amin, professor, Study Chair — Assiut medical school
Locations (1):
- Assiut Medical School, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] El Saman AM. Combined retropubic balloon vaginoplasty and laparoscopic canalization: a novel blend of techniques provides a minimally invasive treatment for cervicovaginal aplasia. Am J Obstet Gynecol. 2009 Sep;201(3):333.e1-5. doi: 10.1016/j.ajog.2009.07.001. PMID 19733291
- [Result] El Saman AM. Endoscopically monitored canalization for treatment of congenital cervical atresia: the least invasive approach. Fertil Steril. 2010 Jun;94(1):313-6. doi: 10.1016/j.fertnstert.2009.02.079. Epub 2009 May 21. PMID 19463998
- [Result] Fedele L, Bianchi S, Frontino G, Berlanda N, Montefusco S, Borruto F. Laparoscopically assisted uterovestibular anastomosis in patients with uterine cervix atresia and vaginal aplasia. Fertil Steril. 2008 Jan;89(1):212-6. doi: 10.1016/j.fertnstert.2007.01.168. Epub 2007 May 4. PMID 17482183
- [Result] Li M, Zhang Z. Laparoscopically assisted biomaterial graft for reconstruction in congenital atresia of vagina and cervix. Fertil Steril. 2013 Dec;100(6):1784-7. doi: 10.1016/j.fertnstert.2013.08.046. Epub 2013 Sep 29. PMID 24083872
- [Result] El Saman AM, Shahin AY, Nasr A, Tawfik RM, Saadeldeen HS, Othman ER, Habib DM, Abdel-Aleem MA. Hybrid septate uterus, coexistence of bicornuate and septate varieties: a genuine report. J Obstet Gynaecol Res. 2012 Nov;38(11):1308-14. doi: 10.1111/j.1447-0756.2012.01866.x. Epub 2012 May 21. PMID 22612567
- [Result] El Saman AM, Nasr A, Tawfik RM, Saadeldeen HS. Mullerian duct anomalies: successful endoscopic management of a hybrid bicornuate/septate variety. J Pediatr Adolesc Gynecol. 2011 Aug;24(4):e89-92. doi: 10.1016/j.jpag.2011.02.013. Epub 2011 Apr 21. PMID 21514191
- [Result] Ozbey H, Morozov D, Morozov DA. Abdominal pain as the presentation of imperforate hymen in a teenage girl. Pediatr Int. 2022 Jan;64(1):e15168. doi: 10.1111/ped.15168. No abstract available. PMID 35438216
- [Result] Rozalska B, Sakata N, Wadstrom T. Staphylococcus aureus fibronectin-binding proteins (FnBPs). Identification of antigenic epitopes using polyclonal antibodies. APMIS. 1994 Feb;102(2):112-8. PMID 8167006